CLINICAL TRIAL: NCT06187233
Title: The Effects of Binaural Beats on Pain, Anxiety, and Procedure Tolerance in Patients Undergoing Colonoscopy Without Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, selim demirci, Clinical physician, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: colonoscopybinaural
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Anxiety State; Patient Satisfaction; Tolerance
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: All elective colonoscopies were performed by an experienced endoscopists who were unaware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- binaural music group (Experimental): The music group listened to music containing binaural beats during the colonoscopy
  Interventions: Other: binaural music
- control (No Intervention): The control group had headphones without sound during the procedure.

INTERVENTIONS:
Other: binaural music — In the binaural music group, an MP3 player and in-ear stereo headphones were provided. Music therapy was applied during the procedure.
  Arms: binaural music group

SUMMARY:
The purpose of this study was to investigate the effect of binaural beats on anxiety, pain and tolerance during colonoscopy without sedation

DETAILED DESCRIPTION:
It is a prospective randomized, controlled, single-blind procedural study included 92 Turkish patients aged 18-70 years old scheduled for colonoscopy regardless of sex or underlying disease. The patients were randomly divided into two groups: the binaural beat music group(n=46) and the control group(n=46). The binaural music group listened to music through headphones during colonoscopy, while the control group had headphones without music. Anxiety levels (VAS-Anxiety scale) were measured both before and after the procedure, and pain levels (VAS-pain) were measured following the procedure. Hemodynamic changes before and after endoscopy , procedure tolerance (using modified gloucester comfort scale), cecal insertion and withdrawal times, polyp detection rate, and patients' experiences related to colonoscopy were recorded. Likert scales were collected as well just after the colonoscopy procedure, indicating satisfaction and willingness to repeat the process.

ELIGIBILITY:
Inclusion Criteria:

- Between 18-70 years old who had scheduled colonoscopy appointments

Exclusion Criteria:

* Anxiety and panic disorders
* Urgent endoscopic intervention
* Advanced dementia
* Hearing problems
* Anatomical or inflammatory disorders in the external ear canals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
VAS-anxiety | immediately before being taken into the procedure room and 5 minutes after the procedure
  The VAS scale, developed by Price et al. (1983), has been employed in recent years to measure patients' subjective experiences of pain and anxiety.This scale utilizes a 10-cm horizontal or vertical line, with the two endpoints representing the minimum and maximum scores for pain and anxiety(0: no pain/no anxiety, 10: the most severe pain/extremely anxious). The colonoscopy nurse recorded patients' pain and anxiety scores by manually marking a 10-cm line. This indicator is a reliable measure for assessing pain and anxiety
VAS-pain | 5 minutes after the procedure
  The VAS scale, developed by Price et al. (1983), has been employed in recent years to measure patients' subjective experiences of pain and anxiety.This scale utilizes a 10-cm horizontal or vertical line, with the two endpoints representing the minimum and maximum scores for pain and anxiety(0: no pain/no anxiety, 10: the most severe pain/extremely anxious). The colonoscopy nurse recorded patients' pain and anxiety scores by manually marking a 10-cm line. This indicator is a reliable measure for assessing pain and anxiety
The Modified Gloucester Comfort Scale | During the procedure
  The endoscopy nurse recorded and analyzed data related to patient comfort, encompassing compliance and tolerance during the procedure, using the Modified Gloucester Comfort Scale.Discomfort, characterized by severe belching, retching, coughing, and non-compliance, was assessed on a scale where the absence of discomfort received a score of 1 point, while extreme discomfort during the procedure was assigned 5 points.

SECONDARY OUTCOMES:
Patient satisfaction | 5 minutes after the procedure
  After the procedure, the patients were asked a series of questions for procedure evaluation (worse than expected, as expected, better than expected) and their willingness to have endoscopy again for their health (no, yes). The binaural music group was asked a three-item question with "yes-not sure-no" responses, inquiring whether the music increased relaxation and if they would like to listen to the same music again during a repeat procedure.
Heart rate | Within 20 minutes pre-procedure and 5 minutes after the procedure
  The comparison of heart rate in the music and control groups
Blood pressure | Within 20 minutes pre-procedure and 5 minutes after the procedure
  The comparison of systolic and diastolic blood pressure in the music and control groups
cecal insertion time(minutes) | during the procedure
  Insertion time, as defined, refers to the duration between the initiation of the colonoscopy procedure and the moment when the endoscope reaches the cecum, with identification of the appendiceal orifice.
withdrawal time (minutes) | during the procedure
  Withdrawal time, as defined, refers to the period between the commencement of withdrawing the colonoscope from the cecum and the complete removal of the colonoscope from the patient.
polyp detection rate | during the procedure
  It will be assessed by recording the encountered polyps during colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: selim demirci, Principal Investigator — clinical physician
Locations (1):
- Abdurrahman Yurtaslan Oncology and Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tani A, Tartarisco G, Vagheggini G, Vaccaro C, Campana S, Tomaiuolo F. Binaural beats reduce feeling of pain and discomfort during colonoscopy procedure in not-sedated patients: A randomized control trial. Complement Ther Clin Pract. 2022 Aug;48:101605. doi: 10.1016/j.ctcp.2022.101605. Epub 2022 May 21. PMID 35623152
- [Result] Isik BK, Esen A, Buyukerkmen B, Kilinc A, Menziletoglu D. Effectiveness of binaural beats in reducing preoperative dental anxiety. Br J Oral Maxillofac Surg. 2017 Jul;55(6):571-574. doi: 10.1016/j.bjoms.2017.02.014. Epub 2017 Mar 18. PMID 28325532
- [Result] Wang MC, Zhang LY, Zhang YL, Zhang YW, Xu XD, Zhang YC. Effect of music in endoscopy procedures: systematic review and meta-analysis of randomized controlled trials. Pain Med. 2014 Oct;15(10):1786-94. doi: 10.1111/pme.12514. Epub 2014 Aug 19. PMID 25139786